CLINICAL TRIAL: NCT06282133
Title: Behavioural Experiments for Intolerance of Uncertainty: A Novel Treatment for Generalized Anxiety Disorder in Adolescents - A Pilot Study
Brief Title: Behavioural Experiments for Generalized Anxiety in Adolescents - Pilot Study
Acronym: EC-II-Ado-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Quebec en Outaouais (Other)
Responsible Party: Principal Investigator, Michel Dugas, Ph.D., Professor of Psychology, Universite du Quebec en Outaouais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1862
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Generalized Anxiety Disorder; Adolescent - Emotional Problem
Keywords: Cognitive-behavioural therapy
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioural Experiments (CBT) (Experimental): Behavioural experiments involve selecting a specific thought to test (for example, "uncertainty makes me incapable of acting") and designing a detailed experiment to challenge this thought.
  Interventions: Behavioral: Behavioural Experiments for Intolerance of Uncertainty

INTERVENTIONS:
Behavioral: Behavioural Experiments for Intolerance of Uncertainty — Behavioural experiments involve selecting a specific thought to test (for example, "uncertainty makes me incapable of acting") and designing a detailed experiment to challenge this thought.
  Other Names: CBT

SUMMARY:
Generalized Anxiety Disorder (GAD) is a chronic condition characterized by excessive and uncontrollable worry and anxiety. In adolescents, this condition can seriously impact their development, academic performance, and social relationships. In Canada, 3 to 4% of the population (between 0.9% and 2.7% among adolescents) suffers from GAD at any given time in their lives. These young individuals experience a reduced quality of life and are at risk for numerous medical conditions, as well as additional psychological issues. Research suggests that both pharmacological and psychological approaches are effective in treating GAD in the short term. However, psychological treatments appear to offer the greatest long-term benefits. There are a number of effective psychological treatments for GAD, most of which fall under cognitive-behavioural therapy (CBT) adapted for this age group.

In the 1990s, a group of Canadian researchers developed a CBT protocol for GAD that included four components. Data from six clinical trials in adults suggest that one of the four components is particularly important for treatment success: exposing oneself to uncertainty rather than avoiding it in daily life. In other words, learning to tolerate and manage uncertainty seems to be the key to reducing worry and anxiety.

Given this discovery, researchers developed a new treatment that exclusively targets intolerance to uncertainty and then adapted it for adolescents: Behavioural Experiments for Intolerance to Uncertainty in Adolescents (EC-IIA). The aim of the current pilot study is to test the effectiveness of EC-IIA in adolescent individuals. A total of 8 participants with a primary diagnosis of GAD will receive EC-IIA and will be evaluated at 4 different times ranging from pre-treatment to a 6-month follow-up. Conditions will be compared in terms of treatment efficacy and mechanisms. Researchers will also examine predictors of change during the 6 months following treatment. The proposed study will produce data on the effectiveness and mechanisms of a treatment for GAD that is less costly, less complex, and easier to disseminate than currently available treatments.

ELIGIBILITY:
Inclusion Criteria:

Adolescents aged between 14 and 18 years; 2) primary diagnosis of Generalized Anxiety Disorder (GAD); 3) no change in type or dose of medication in the 4 to 12 weeks preceding entry into the study (4 weeks for benzodiazepines, 12 weeks for antidepressants, hypnotics, and psychostimulants); 4) willingness to maintain stable medication status during participation in the study; 5) absence of consumption of herbal products known to have effects on the central nervous system in the 2 weeks preceding entry into the study; 6) absence of evidence of suicidal intent (based on clinical judgment); 7) absence of evidence of current substance use, current or past schizophrenia, bipolar disorder, or organic mental disorder; 8) absence of current participation in other clinical trials (i.e., psychotherapeutic services); 9) absence of concurrent psychotherapy during the trial treatment phase; 10) absence of evidence of anxiety symptoms due to a general medical condition based on clinical judgment (e.g., clinical hyperthyroidism, hypoglycemia, anemia).

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-5) | 10 weeks
  Structured diagnostic interview

SECONDARY OUTCOMES:
Worry and Anxiety Questionnaire (WAQ) | 10 weeks
  Self-report questionnaire
Penn State Worry Questionnaire (PSWQ) | 10 weeks
  Self-report questionnaire
Beck Anxiety Inventory (BAI) | 10 weeks
  Self-report questionnaire
Beck Depression Inventory-II (BDI-II) | 10 weeks
  Self-report questionnaire

OTHER OUTCOMES:
Intolerance of Uncertainty Scale (IUS) | 10 weeks
  Self-report questionnaire
Safety Behaviors Questionnaire (SBQ) | 10 weeks
  Self-report questionnaire
Treatment Acceptance and Adherence Scale (TAAS) | 3 weeks
  Self-report questionnaire
Working Alliance Inventory (WAI) | 3 weeks
  Self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michel J. Dugas, Ph.D., Principal Investigator — Universite du Quebec en Outaouais
Locations (1):
- Universite du Quebec en Outaouais, Gatineau, Quebec, Canada